CLINICAL TRIAL: NCT02043405
Title: Weight Loss and/or Exercise Training to Discover Muscle Lipids Related to Insulin Sensitivity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-1551; UL1TR001082 (NIH)
Record Dates: First submitted 2014-01-16; First posted 2014-01-23 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Diabetes; Pre-diabetes
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Training and Weight Loss Intervention (Experimental): Combination weight loss/exercise training, on insulin sensitivity, muscle lipid composition and localization in skeletal muscle.
  Interventions: Behavioral: Weight loss and exercise training intervention
- 4 Month Weight Loss Only Intervention (Active Comparator): Use exercise training and weight loss as separate interventions in obese subjects with and without pre-diabetes.
  Interventions: Behavioral: Weight loss Only Intervention

INTERVENTIONS:
Behavioral: Weight loss and exercise training intervention — Combined weight loss and exercise training intervention
  Arms: Exercise Training and Weight Loss Intervention
Behavioral: Weight loss Only Intervention — Weight loss Only Intervention
  Arms: 4 Month Weight Loss Only Intervention

SUMMARY:
The investigators will use exercise training and weight loss to discover localized lipid species related to diabetes risk in people.

ELIGIBILITY:
Inclusion Criteria:

* Obese men and women with pre-diabetes; (BMI 30-40 kg/m2)
* Ages ranging from 30-60 years old;
* Individuals with:

  * impaired fasting glucose (IFG), (between 100-125mg/dl, with post-prandial glucose (<140 mg/dl 2 hrs after 75g OGTT)
  * impaired glucose tolerance (IGT), (normal fasting glucose <100mg/dl, with post-prandial glucose (>140 mg/dl 2 hrs after 75g OGTT)
  * a combination of the two (IFG/IGT) (both impaired fasting glucose (100-125mg/dl), and impaired glucose tolerance (>140 mg/dl 2 hrs after 75g OGTT), will be verified using oral glucose tolerance testing at initial screening, and
* Sedentary (<2 hours/week of planned physical activity).

To increase generalizability, and because each subject serves as their own control, women will be enrolled regardless of menopausal status, use of hormone replacement therapy and oral contraceptives.

Exclusion Criteria:

* Regular exercise more than 2 hours/week,
* medications that could affect glucose,
* lipid metabolism,
* thyroid disease,
* history of lung disease,
* pregnancy,
* active cigarette smoking or exposure to second hand smoke, and
* Severe plasma lipid disorders.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08-03 (Actual); Study Completion 2015-08-03 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity | baseline and 3 months
  Change in insulin sensitivity measured before and after the 3 month weight loss and exercise training intervention

SECONDARY OUTCOMES:
Change in membrane localized diacylglycerol species | baseline and 3 months
  Change in concentration of membrane and cytosolic diacylglycerol species before and after the intervention. Diacylglycerol is a lipid known to be related to insulin resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Bergman, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

REFERENCES:
- [Derived] Zarini S, Zemski Berry KA, Kahn DE, Garfield A, Perreault L, Kerege A, Bergman BC. Deoxysphingolipids: Atypical Skeletal Muscle Lipids Related to Insulin Resistance in Humans That Decrease Insulin Sensitivity In Vitro. Diabetes. 2023 Jul 1;72(7):884-897. doi: 10.2337/db22-1018. PMID 37186949